CLINICAL TRIAL: NCT02274571
Title: Tissue Selective Estrogen Complex to Prevent Metabolic Dysfunction in Women
Brief Title: Raising Insulin Sensitivity in Post Menopause
Acronym: RISE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 2014-039
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): TSEC (Duavee™, combination of CE and BZA)
  Interventions: Drug: TSEC (Tissue-selective estrogen complexes); Other: Placebo
- Placebo (Placebo Comparator): Non active comparator
  Interventions: Drug: TSEC (Tissue-selective estrogen complexes); Other: Placebo

INTERVENTIONS:
Drug: TSEC (Tissue-selective estrogen complexes) — Duavee™, combination of CE(conjugated equine estrogens) and BZA (bazedoxifene)
  Other Names: Duavee™
Other: Placebo — non active

SUMMARY:
The purpose of this study is to find out if a novel drug approved by the Food and Drug Administration [Duavee™, Pfizer, Inc] for treatment of postmenopausal symptoms (vaginal dryness and hot flashes) and prevention of osteoporosis also improves insulin sensitivity by decreasing body fat especially in your liver.

DUAVEE™ (Conjugated Estrogens/Bazedoxifene) is a new prescription medicine that contains a mixture of estrogen (the main female hormone made by the ovaries) and bazedoxifene, which is FDA approved. For over 60 years, estrogens have been used as hormonal treatments to help manage hot flashes and help prevent postmenopausal bone loss. But in the treatment of postmenopausal women, the use of estrogens alone can increase the risk of developing cancer of the uterus. So estrogens have been traditionally paired with a progestin to decrease the risk of hyperplasia (the thickening of the lining of the uterus), which can be a precursor to cancer. DUAVEE™ uses bazedoxifene, a selective estrogen receptor modulator (SERM), in place of a progestin to help protect the uterus against thickening of the uterus that may result from estrogens alone.

In this study, you will get either DUAVEE™ or the placebo (a "dummy pill" that may look like medicine but contains no active medication) first and then switch to the other pill.

DETAILED DESCRIPTION:
This study involves a screening process to see if you are eligible to participate followed by two 8-week treatment periods separated by an 8-week washout period. The two 8-week treatments will be with:

1. 8 weeks of treatment with TSEC (Duavee™, combination of CE and BZA)
2. 8 weeks of treatment with a "dummy pill" (Placebo) The order of these 2 8-week treatment periods will be decided by chance (coin flip).

   STUDY VISITS (11 VISITS in total) If you participate in this study, after referral from the Baton Rouge General Obstetrics and Gynecology Physicians, you will complete 1 screening visit at Pennington Biomedical Research Center to determine your eligibility. If you are eligible and enrolled in the study, you will complete an additional 10 visits (8 brief visits and 2 overnight inpatient stays).

   Please note all times provided for procedures and the total times for each clinic visit are approximations and may vary depending on circumstances.

   SCREENING VISIT (1 visit, approximately 1.5 hours, fasting):

   Please do not drink any food or water for 10 hours before this appointment.

   Participants are asked to report to the Pennington clinic fasting. After a detailed explanation of the whole study by a coordinator, if you agree to the procedures by signing a consent form, you will have:
   1. Your height and body weight measured.
   2. You will then have an ECG (electrocardiogram) to measure your heart rate and rhythm.
   3. Your blood pressure will be measured.
   4. A blood sample (<1 teaspoon) and urine will be collected to assess your general health.
   5. You will have a medical history and physical examination.

   If fully eligible according to the data collected during the screening visit, you will be called to set up a second visit to provide you with the medication or the dummy pill.

   VISIT 2 (30 minutes):

   You will come to the Pennington to pick up your drug supply (real medication or dummy pill) and meet with a nurse or a study coordinator to give you instructions on when and how to take your pill once a day.

   VISITS 3-5 (30 minutes each):

   At week 1, 3, and 5 of your 8-week treatment period, you will come to our outpatient clinic to measure your weight, blood pressure and pulse, collect some feedback on your health and check your medication compliance as well as distribute new medications.

   VISIT 6 (24 hours at our inpatient unit):

   You will be admitted to our inpatient unit at 4pm (not fasted) for measures of:
   1. Total body fat by DXA
   2. Abdominal visceral fat by Magnetic Resonance Imaging (MRI)
   3. Fat in your liver and muscle by Magnetic Resonance Spectroscopy (MRS) You will then receive a standard dinner at ~7pm and will be ask to switch off the light in your bedroom at ~10pm

   The next morning investigators will wake you up at ~4.45am to start an IV line and start a 8-hour procedure (Euglycemic Clamp) to measure how your body responds to insulin. You will be discharged from the inpatient unit between 2 and 3 pm after being fed a lunch.

   Visit 1 is Screening; Visit 2/7 is Wk0/17; Visit 3/8 is Wk1/18; Visit 4/9 is Wk3/20; Visit 5/10 is Wk5/22 and Visit 6/11 is Wk8/25

   ECG: Screening Vital Signs, Height, Weight, Waist & Hip Measurements: Screening, Visit 3, Visit 4, Visit 5 & Visit 6

   Fasting Blood & Urine Sample: Screening and Visit 6

   Medical History & Physical Exam + Questionnaire Barriers: Screening

   Pick up pills/receive instructions: Visit 2, Visit 3, Visit 4, & Visit 5

   Health Status/Medication Compliance Visit 3, Visit 4 & Visit 5

   Admittance to Inpatient Unit: Visit 6

   Body Composition (DXA): Visit 6

   Body Composition (MRI): Visit 6

   Liver/Muscle Fat (MRS): Visit 6

   Euglycemic Clamp with biopsies: Visit 6

   Eight weeks later (during which you will not take any pill), you will start the same sequence of visits (VISITS 7-11) as shown above for Visits 2-6 but this time with the other pill.

   DESCRIPTION OF PROCEDURES

   Euglycemic IV clamp (8 hours):

   This procedure measures how the body responds to insulin. Insulin is normally produced by your body during meals and helps your body use sugar. There will be 2 IV lines, one in your arm and one in your hand on the opposite side. Approximately 30 minutes after the IV lines are inserted; investigators will perform a fat biopsy to sample fat cells beneath the skin of your stomach area. Then, a muscle biopsy will be obtained to sample muscle cells beneath the skin of your thigh. Small amounts of glucose and insulin will be infused into your arm. Your blood sugar level will be checked every 5-10 minutes from the IV in your hand to determine how much glucose you should have to keep your blood sugar at a normal level. Your hand will be placed inside a warming box to increase skin temperature to about 105 degrees Fahrenheit. The temperature will be warm, but not uncomfortable. During your IV procedure, a small amount of your own blood (less than 1 teaspoon) will immediately be returned into your vein through the IV after each specimen is collected

   Three times during the 8-hour procedure, investigators will place a clear plastic hood, through which fresh air flows, over your head to measure how many calories your body burns. This measure will last 40 minutes each time. Your urine will be collected throughout the test in a urine jug (at the end of the test or in 2 collections if necessary).

   Fat biopsy (about 30 minutes):

   This procedure is used to sample fat cells from underneath the abdominal skin after cleansing the skin with iodine and using a local anesthetic. After cleansing the area, the doctor or Nurse Practitioner will make a small incision in the skin and introduce a needle under the skin to remove fat cells. About 1 gram (less than half a teaspoon size) of fat will be removed. After the biopsy is completed, the skin will be held closed with a sterile adhesive bandage; an antibiotic ointment will be applied.

   Risks: Fat Biopsy: Mild to severe pain, soreness, and bruising, and a small scar are common risks. There is a small risk of a hematoma (collection of blood in the tissue) or infection at the biopsy site. Sterile technique will be used to minimize these risks and the biopsy site will be monitored closely.

   Muscle Biopsy (about 30 minutes):

   This procedure is used to sample muscle cells from underneath the skin of the leg. After cleaning the skin with iodine and using a local anesthetic, the doctor or nurse practitioner will make a small incision in the skin and introduce a needle under the skin to remove muscle cells. About 200-750 milligrams (less than a teaspoon size) of muscle will be removed. After the biopsy is completed, the skin will be held closed with a sterile adhesive bandage and an antibiotic ointment will be applied.

   Risks: Muscle Biopsy: Mild to severe pain, soreness, bruising, and a small scar are common risks. A hematoma (collection of blood in the tissue) may occur. There is a slight risk that a superficial nerve may be cut; the nerve may heal, or it may result in a permanent loss of sensation in the skin at the biopsy site.

   DXA - Whole Body Scan (~4 minutes):

   This scan measures the amount of bone, muscle, and fat in your body. The scan will be performed using a whole-body scanner. You will be required to wear a hospital gown, to remove all metal-containing objects from your body, and to lie down on the table. A scanner emitting low energy X-rays and a detector will pass along your body. You will be asked to remain completely still while the scan is in progress. The scan takes less than four minutes. This scan is for research purposes only and not for diagnostic treatment.

   MRI Abdomen (30 minutes):

   This scan measures the amount of fat in your abdomen. You will change into a hospital gown and remove all objects containing metal from your body. You will lie on your back on the scanner table with your arms above your head. A large coil will be placed around your upper abdomen. You will then be moved into the magnet and will be instructed to hold your breath 4-5 times (once for six seconds, once for 13 seconds, and 2-3 times for about 18 seconds after the upper abdominal scans are completed, you will be moved up on the table, and the coil will be placed over your lower abdomen. The same scans will be acquired over this area with the same 4-5 breath holds. The total scan time for this procedure is approximately 30 minutes. During the scan, you will hear loud tapping noises. You will be given headphones for protection from the scanner noise and can listen to music during the scan if desired. You will also be given a call button should you need the MRI Technician during the exam. This scan is for research purposes only and not for diagnostic treatment.

   MRS IHL (Intrahepatic lipid) (20-30 minutes):

   This scan measures the amount of fat in your liver. You will change into a hospital gown and remove all objects containing metal from your body. You will be placed on the scanner table head first and on your stomach. The table will move you into the magnet where data will be obtained. The scan will last for approximately 20-30 minutes. During the scan, you will hear loud tapping noises. You will be given head phones for protection from the scanner noise and can listen to music during the scan if desired. You will also be given a call button should you need the MRI tech during the exam. This scan is for research purposes only and not for diagnostic treatment.

   MRS IMCL (Intramyocellular lipid) (60 minutes):

   This scan measures the amount of fat in your muscle fibers. You will change into a hospital gown and remove all objects containing metal from your body. You will lie on your back on the scanner table with the right leg in a special coil. The top part of the coil will then be placed over your calf. Cushions will be inserted around the calf to help keep the leg as still as possible. The table will then move you into the scanner where a series of several scans will be obtained. The entire procedure will last approximately 60 minutes. During the scan, you will hear loud tapping noises. You will be given head phones for protection from the scanner noise and can listen to music during the scan if desired. You will also be given a call button should you need the MRI tech during the exam. This scan is for research purposes only and not for diagnostic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (<5y post last period)
* Age between 50-60y
* Symptomatic (hot flashes, vaginal dryness) or asymptomatic
* BMI 30-40 kg/m2
* Normal mammogram past 12 months
* Physician clearance (Ob/Gyn or PBRC)

Exclusion Criteria:

* Amenorrhea other causes (excess androgen)
* Diabetes mellitus
* Medications: diabetes, antidepressant uncontrolled depression (2 months stability on SSRIs are fine), antipsychotics, oral steroids, weight loss drugs
* Tricyclic antidepressants (TCAs)
* ≤ 3 month washout of birth control pill, estrogen, and/or progestin
* Hysterectomy (total or partial)
* Contraindications to estrogen treatment
* Unable or unwilling to do an MRS

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 269 applied to participate. 82 completed a web base screening. 18 screened in the clinic. 10 were ineligible and 8 enrolled and were randomized and completed the study.
Pre-assignment Details: the 10 ineligible were 5 BMI out of range. 2 > 5 year post menopause. 1 because of medication. 1 for medical condition and 1 failed to return to clinic.
Groups:
- TSEC (Duavee™, Combination of CE and BZA), Then Placebo: Participants received TSEC 0.45/20 mg per day each for an 8-week treatment period, then after an 8-week washout, participants received Placebo tablet (matching TSEC 0.45/20 mg per day each for an 8-week treatment period).
- Placebo, Then TSEC (Duavee™, Combination of CE and BZA): Participants received Placebo tablet (matching TSEC 0.45/20 mg per day each for an 8-week treatment period), then after an 8-week washout, participants received TSEC 0.45/20 mg per day each for an 8-week treatment period.
Period: Overall Study
Arm/Group | TSEC (Duavee™, Combination of CE and BZA), Then Placebo | Placebo, Then TSEC (Duavee™, Combination of CE and BZA)
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Female Participants: This study involves a screening process to see if you are eligible to participate followed by two 8-week treatment periods separated by an 8-week washout period. The two 8-week treatments will be with:
  8 weeks of treatment with TSEC (Duavee™, combination of CE and BZA) 8 weeks of treatment with a "dummy pill" (Placebo) The order of these 2 8-week treatment periods will be decided by chance (coin flip).
Arm/Group | Enrolled Female Participants
Number analyzed (Participants) | 8
Age, Customized [Number; unit: years]
  Age 50-60 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Effect of CE/BZA (TSEC) on Body Composition
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Groups:
- Placebo: Participants received TSEC 0.45/20 mg per day each for an 8-week treatment period.
  Two 8-week treatment periods separated by an 8-week washout period. The two 8-week treatments will be with:
  8 weeks of treatment with TSEC (Duavee™, combination of CE and BZA) 8 weeks of treatment with a "dummy pill" (Placebo) The order of these 2 8-week treatment periods will be decided by chance (coin flip).
- TSEC (Duavee™, Combination of CE and BZA): Participants received Placebo tablet (matching TSEC 0.45/20 mg per day each for an 8-week treatment period)
  Two 8-week treatment periods separated by an 8-week washout period. The two 8-week treatments will be with:
  8 weeks of treatment with TSEC (Duavee™, combination of CE and BZA) 8 weeks of treatment with a "dummy pill" (Placebo) The order of these 2 8-week treatment periods will be decided by chance (coin flip).
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
Kilograms
  Weight | 91.3 (6.8) | 90.6 (7.2)
  Fat Mass | 45.5 (4.6) | 45.7 (4.0)
  Fat-free Mass | 46.0 (3.5) | 45.5 (4.0)

2. Primary Outcome: Effect of CE/BZA (TSEC) on Ectopic Fat - 1H-MRS, Proton Magnetic Resonance Spectroscopy
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
Percent
  Intrahepatic Lipid (IHL) | 9.00 (13.9) | 8.06 (9.14)
  Soleus intramyocellular lipid (IMCL) | 0.29 (0.27) | 0.36 (0.47)
  Soleus extramyocellular lipid (EMCL) | 0.32 (0.28) | 0.43 (0.45)
  Tibialis anterior intramyocellular lipid (IMCL) | 0.33 (0.23) | 0.69 (0.50)
  Tibialis anterior extramyocellular lipid (EMCL) | 1.87 (1.60) | 4.13 (6.06)

3. Primary Outcome: Effect of CE/BZA (TSEC) on Abdominal Fat Cell Size (by Biopsy)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
Percent
  Small Fat Cells | 66.4 (8.7) | 66.0 (5.5)
  Large Fat Cells | 33.6 (8.7) | 34.0 (5.5)

4. Primary Outcome: Effect of CE/BZA (TSEC) on Body Mass Index
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kilograms per meter squared
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
kilograms per meter squared | 36.6 (2.7) | 36.4 (2.9)

5. Primary Outcome: Effect of CE/BZA (TSEC) on Percent Body Fat
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of total body weight
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
percentage of total body weight | 50.9 (2.5) | 51.4 (1.9)

6. Primary Outcome: Effect of CE/BZA (TSEC) on Fat Cell Ratio (Small/Large)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
ratio | 2.19 (1.00) | 2.00 (0.45)

7. Primary Outcome: Effect of CE/BZA (TSEC) on Mean Fat Cell Size
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: um^3 (x10^6)
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
um^3 (x10^6) | 1.35 (0.4) | 1.6 (0.4)

8. Secondary Outcome: Effect of CE/BZA (TSEC) on Fasting Labs
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Milligrams/deciliter
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
Milligrams/deciliter
  Glucose | 105 (4) | 102 (4)
  Total cholesterol | 179 (34) | 187 (32)
  Triglycerides | 138 (75) | 156 (73)
  HDL-cholesterol | 51 (11) | 57 (14)
  LDL-cholesterol | 100 (24) | 99 (20)

9. Secondary Outcome: Effect of CE/BZA on Insulin Sensitivity (by Hyperinsulinemic-Euglycemic Clamp)
Description: Low-Dose Insulin [20 mIU/min/m2 ], High-Dose Insulin [120 mIU/min/m2 ]
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/min [FFM+17.7]
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
mg/min [FFM+17.7]
  Basal SGO | 2.83 (0.41) | 2.68 (0.32)
  GDR at Low-Dose Insulin | 2.48 (0.91) | 2.55 (1.04)
  GDR at High-Dose Insulin | 11.99 (4.49) | 11.68 (4.23)

10. Secondary Outcome: Effect of CE/BZA (TSEC) on Insulin Sensitivity (by Hyperinsulinemic-Euglycemic Clamp) on FFA
Description: Low-Dose Insulin [20 mIU/min/m2 ] High-Dose Insulin [120 mIU/min/m2 ]
Time Frame: 8 weeks
Population: No data reported for FFA for High-Dose Insulin
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
mmol/L
  Free Fatty Acids (FFA) at Low-Dose Insulin | 0.13 (0.05) | 0.13 (0.05)
  Free Fatty Acids (FFA) at High-Dose Insulin | 0 (0) | 0 (0)

11. Secondary Outcome: Effect of CE/BZA (TSEC) on Resting Metabolic Rate & Substrate Oxidation (by Indirect Calorimetry)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
kcal/day
  Resting Metabolic Rate (RMR) on Basal | 1410 (126) | 1471 (161)
  Resting Metabolic Rate (RMR) on Low-Dose Insulin | 1379 (94) | 1378 (137)
  Resting Metabolic Rate (RMR) on High-Dose Insulin | 1516 (113) | 1576 (83)

12. Secondary Outcome: Effect of CE/BZA (TSEC) on Resting Metabolic Rate & Substrate Oxidation (by Indirect Calorimetry)
Description: Low-Dose Insulin [20 mIU/min/m2 ], High-Dose Insulin [120 mIU/min/m2 ]
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/min/[FFM+17.7]
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
mg/min/[FFM+17.7]
  Carbohydrate Oxidation at Basal | 1.2 (0.1) | 1.0 (0.1)
  Carbohydrate Storage at Basal | 1.6 (0.3) | 1.6 (0.3)
  Carbohydrate Oxidation at Low-Dose | 1.6 (0.1) | 1.3 (0.1)
  Carbohydrate Storage at Low-dose | 0.9 (0.3) | 1.2 (0.3)
  Carbohydrate Oxidation at High-Dose | 2.7 (0.3) | 2.7 (0.3)
  Carbohydrate Storage at High-Dose | 9.3 (1.4) | 9.0 (1.4)

13. Secondary Outcome: Effect of CE/BZA (TSEC) on Resting Metabolic Rate & Substrate Oxidation (by Indirect Calorimetry)
Description: Low-Dose Insulin [20 mIU/min/m2 ], High-Dose Insulin [120 mIU/min/m2 ]
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
unitless
  Respiratory Quotient (RQ) at Basal | 0.81 (0.03) | 0.80 (0.03)
  Respiratory Quotient (RQ) at Low-Dose | 0.85 (0.04) | 0.83 (0.03)
  Respiratory Quotient (RQ) at Hight-Dose | 0.92 (0.05) | 0.91 (0.06)

14. Secondary Outcome: Effect of CE/BZA (TSEC) on Fasting Insulin
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
uU/mL | 16.6 (2.8) | 15.7 (2.8)

15. Secondary Outcome: Effect of CE/BZA (TSEC) on Fasting Free Fatty Acids
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
mmol/L | 0.72 (0.06) | 0.78 (0.06)

16. Secondary Outcome: Effect of CE/BZA on Insulin Sensitivity (by Hyperinsulinemic-Euglycemic Clamp) on Glucose
Description: Low-Dose Insulin [ 20 mIU/min/m2 ]
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
mg/dL
  Low-Dose Glucose | 90 (1) | 88 (1)
  High-Dose Glucose | 97 (3) | 95 (3)

17. Secondary Outcome: Effect of CE/BZA (TSEC) on Insulin Sensitivity (by Hyperinsulinemic-Euglycemic Clamp) on Insulin
Description: Low-Dose Insulin [20 mIU/min/m2 ] High-Dose Insulin [120 mIU/min/m2 ]
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
Number analyzed (Participants) | 8 | 8
uU/mL
  Insulin at Low-Dose Insulin | 37.8 (2.4) | 34.8 (2.4)
  Insulin at High-Dose Insulin | 250.8 (19.3) | 259.8 (19.3)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: For reporting AE and SAE, all subject population was used.
Groups:
- Placebo: Participants received Placebo tablet (matching TSEC 0.45/20 mg per day each for an 8-week treatment period), then after an 8-week washout, participants received TSEC 0.45/20 mg per day each for an 8-week treatment period
- TSEC (Duavee™, Combination of CE and BZA): Participants received TSEC 0.45/20 mg per day each for an 8-week treatment period, then after an 8-week washout, participants received Placebo tablet (matching TSEC 0.45/20 mg per day each for an 8-week treatment period)
Arm/Group | Placebo | TSEC (Duavee™, Combination of CE and BZA)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | TSEC (Duavee™, Combination of CE and BZA) (N=8)
Neuropsychiatric (Psychiatric disorders) | 1 (1) | 1 (2)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Hematologic/oncologic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — bruising to (R) elbow caused by fall
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Genitourinary (Renal and urinary disorders) | 2 (2) | 0 (0)
Neurological (Nervous system disorders) | 0 (0) | 1 (1)
Oral Complaints (General disorders) | 0 (0) | 1 (1)
Nonspecific (General disorders) | 1 (1) | 0 (0)
Special Senses (General disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT02274571/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT02274571/ICF_001.pdf